CLINICAL TRIAL: NCT01179893
Title: A Randomized Trial of Plasma Exchange vs. IVIG in the Treatment of Myasthenia Gravis
Brief Title: Intravenous Immunoglobulin and Plasma Exchange in Myasthenia Gravis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Grifols Therapeutics LLC (Industry)
Responsible Party: Vera Bril, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0280-B
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Myasthenia Gravid
Keywords: Myasthenia Gravis; IVIG; PLEX
MeSH Terms: conditions — Myasthenia Gravis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVIG (Active Comparator): Intravenous Immunoglobulin, 2G/Kg, infused over 2 days in the Medical Day Unit of the University Health Network
  Interventions: Biological: IVIG
- PLEX (Experimental): Patients received one plasma volume plasma exchanges with 5% albumin replacement fluid. Five plasma exchange procedures occurred every second day with breaks over the weekend allowed. Patients treated in the apheresis units at the University Health Network.
  Interventions: Procedure: PLEX

INTERVENTIONS:
Biological: IVIG — Intravenous immunoglobulin
  Arms: IVIG
Procedure: PLEX — Plasma exchange: removal of pathogenic antibodies and constituents and replacement with albumin.
  Arms: PLEX

SUMMARY:
Immunomodulation is effective in treating patients with myasthenia gravis (MG), but prior studies have not adequately defined if plasma exchange (PLEX) in superior to intravenous immunoglobulin (IVIG) in the treatment of myasthenia gravis. This study aimed to determine if PLEX was superior to IVIG in the treatment of patients with myasthenia gravis.

Patients with MG requiring immunomodulation are randomized to IVIG or PLEX and treated with a full course of immunomodulation. The quantitative myasthenia gravis score (QMGS) will be evaluated as the primary efficacy parameter at day 14 to determine if PLEX is superior to IVIG.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* diagnosis of moderate-severe MG (defined as a Quantitative Myasthenia Gravis Score QMGS >10.5)
* worsening weakness requiring a change in therapy judged by a neuromuscular expert

Exclusion Criteria:

* Worsening weakness secondary to concurrent medications (e.g. Aminoglycosides)
* Worsening weakness secondary to infection
* Change in corticosteroid dosage in the 2 weeks prior to screening
* Other disorders causing weakness or fatigue
* Known absolute IgA deficiency (risk of anaphylactic reaction to IVIG)
* History of anaphylaxis or severe systemic response to IVIG or albumin
* Pregnancy or breastfeeding
* Active renal failure precluding volume of IVIG (risk of volume overload with IVIG) as judged by the investigators
* Clinically significant cardiac disease precluding IVIG volume as judged by the investigators
* Known hyperviscosity or hypercoaguable state (risk of stroke with IVIG)
* Known coagulopathy with bleeding
* On another current study medication or protocol within 4 weeks of screening
* Patients with known refractory status to either IVIG or PLEX
* Poorly controlled or severe hypertension (exacerbation by IVIG)
* Patient refuses treatment with either IVIG or PLEX
* Patient refuses follow-up with electrophysiological studies
* Patient unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in Quantitative Myasthenia Gravis Score (QMGS) from baseline to day 14 after treatment | QMGS at day 14, and patients followed to day 60
  QMGS is a validated clinical measure of myasthenia gravis ranging from 0 points (no myasthenic weakness) to a maximum of 39 points, with a defined change of 3.4 units required for clinical significance.

SECONDARY OUTCOMES:
QMGS Score change at days 21 and 28 from start of treatment. | 28 days
  Change in QMGS with time to see if effect ad day 14 is sustained.
Post intervention status | Day 14, 21 and 28
  Categorical scale of improvement, worsening, or no change for myasthenia gravis.
Single fiber electromyography: jitter, percent abnormal pair, percent blocking | Days 14 and 28 compared to baseline
  Electrophysiological assessment of neuromuscular transmission.
Repetitive Nerve stimulation studies | Days 14 and 28
  Assessment of decrement
Acetylcholine Receptor Antibody titers | Day 28 (if positive at baseline)
  Laboratory assay of pathogenic antibody
AntiMUSK antibody | Day 28 (if positive at baseline)
  Laboratory measure of pathogenic antibody
Need for ICU admission, ventilation, intubation | 60 days
  Myasthenic deterioration and crisis
Hospitalization | 60 days
  Myasthenic deterioration and crisis
Need for additional myasthenic treatment | Day 60
  Myasthenic deterioration or crisis

CONTACTS AND LOCATIONS:
Overall Officials: Vera Bril, BSc, MD, FRCPC, Principal Investigator — University Health Network, Toronto; David Barth, MD, Principal Investigator — University Heatlh Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Zinman L, Ng E, Bril V. IV immunoglobulin in patients with myasthenia gravis: a randomized controlled trial. Neurology. 2007 Mar 13;68(11):837-41. doi: 10.1212/01.wnl.0000256698.69121.45. PMID 17353471